CLINICAL TRIAL: NCT06978504
Title: What is the Impact of Genetic Polymorphisms and DASH Diet On Weight Loss Progression In Climacteric Women With Metabolic Syndrome?
Brief Title: Impact of Genetic Polymorphisms And DASH Diet On Weight Loss Progression In Climacteric Women With Metabolic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrindo Ideais Research Center (Network)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79705724.2.0000.5257
Record Dates: First submitted 2025-04-26; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Nutrition; Metabolic Syndrome; Obesity; Weight Loss; Genetic Polymorphisms
Keywords: Dash; Nutrition; Weight Loss; metabolic Syndrome; genetic polymorphisms
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Weight Loss | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): 30 menopausal women aged between 40 and 60 years who are obese (BMI > 30) and diagnosed with metabolic syndrome. Volunteers will have in-person and online consultations with a nutritionist every 15 days for 3 months to assess their previous habitual food intake and their nutritional adherence to DASH Diet.
  Interventions: Other: DASH diet

INTERVENTIONS:
Other: DASH diet — Prospective, single-arm, unblinded clinical trial lasting 90 days. The study population will consist of menopausal women aged between 40 and 60 years who are obese (BMI > 30) and diagnosed with metabolic syndrome. Volunteers will have an in-person consultation with a nutritionist at t0 to assess their previous habitual food intake and will receive a DASH diet. To minimize losses during the study, in-person consultations with a nutritionist will be held at t0, t30, t60, t90 and online consultations (teleconsultation) at t15, t45 and t75 to answer a questionnaire to assess nutritional adherence that will be applied by the nutritionist. Saliva samples will be collected for genetic panel analysis only at t90. Serum samples for analysis of lipid profile, blood glucose, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), follicle stimulating hormone (FSH), C-reactive protein (CRP) and tumor necrosis factor (TNF) and profile of medications used will be collected at t0 and t90.

SUMMARY:
Metabolic syndrome is a multifactorial inflammatory condition that is very prevalent in overweight women with type 2 diabetes. However, there seems to be great benefit in changing lifestyle and dietary patterns in the treatment of this condition. Currently, few studies have shown the effect of a Dietary Approach to Stop Hypertension (DASH) diet in postmenopausal women with metabolic syndrome and the influence of genetic polymorphisms of the fat mass and obesity-associated protein (FTO) and beta-2 adrenergic receptor (ADRB2) genes on inflammatory markers and improvement of laboratory indicators in these patients. This study aims to analyze the interaction of polymorphisms in the ADRB2 and FTO genes and the DASH diet on anthropometric indicators and laboratory tests in patients with metabolic syndrome in the city of Rio de Janeiro. For this purpose, laboratory tests and anthropometric data will be collected in a prospective study with women aged between 40 and 60 years.

DETAILED DESCRIPTION:
Prospective, single-arm, unblinded clinical trial lasting 90 days. The study population will consist of menopausal women aged between 40 and 60 years who are obese (BMI > 30) and diagnosed with metabolic syndrome. Volunteers will have an in-person consultation with a nutritionist at t0 to assess their previous habitual food intake and will receive a DASH diet. To minimize losses during the study, in-person consultations with a nutritionist will be held at t0, t30, t60, t90, and online consultations (teleconsultation) at t15, t45 and t75 to answer a questionnaire to assess nutritional adherence that the nutritionist will apply. Saliva samples will be collected for genetic panel analysis only at t90. Serum samples for analysis of lipid profile, blood glucose, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), follicle stimulating hormone (FSH), C-reactive protein (CRP) and tumor necrosis factor (TNF) and profile of medications used will be collected at t0 and t90.

Only one nutritionist will make the dietary prescription to maintain the standardization of the research. The diets will be previously calculated, varying from 100 to 100 kcal (1400 to 2600 kcal) based on the patients' total energy value (TEV). The isocaloric, balanced, and individualized diet will be calculated according to the resting metabolic rate (RMR) obtained by the prediction equation and multiplied by the corresponding activity factor to obtain the TEV. The DASH eating plan will consist of fruits, vegetables, legumes, whole grains, and low-fat dairy products. White meat will be prioritized over red meat, seeds and oilseeds will be included, and sweets and foods rich in sodium will be limited.

Dietary assessment will be performed using periodic dietary record forms (24-hour records) for three non-consecutive days, two typical days, and one atypical day, to analyze the participants' eating habits before the dietary intervention. The participants will complete periodic records at seven points before the intervention begins at t15, t30, t45, t60, t75, and at the end of the 90-day study. The nutritionist will review all forms to check for any missing information (number of meals, added sugar, spoon size, quantity consumed, and type of preparation) and notes that could raise questions later (few items recorded, unknown foods, errors in household measurements, and absence of any meal).

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of menopausal women aged between 40 to 60 years old
* Obese (BMI > 30) with a diagnosis of MS.

The inclusion criteria are the presence of at least 3 of the 5 criteria* for MS, which include:

* Abnormal waist circumference values (≥89 cm in women)
* SBP ≥120 mm Hg and DBP ≥80 mm Hg) or diagnosis of hypertension
* Fasting blood glucose equal to or greater than 100 mg/dL or diagnosis of DM2
* HDL-c less than 50 mg/dL in women
* Triglycerides ≥150 mg/dL.

Exclusion Criteria:

* Patients with a BMI <25 kg/m2

The following chronic diseases will not be eligible:

* Active cancer
* Active tuberculosis
* Psychiatric illnesses
* Multiple sclerosis
* Severe nephropathy
* Advanced stages of Paget's disease.

These chronic conditions could interfere with the results of this study, especially adherence to diet and weight loss. Patients who do not complete all stages of the study, who are not adhering to the intervention or who present any complication that interferes with the results of the study will be excluded from the study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Systolic and Diastolic blood pressure in mmHg | Baseline
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken using an Omron IntelliSense® Blood Pressure Monitor and an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals, and the average of the three measurements will be used.
Systolic and Diastolic blood pressure in mmHg | 30 days
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken using an Omron IntelliSense® Blood Pressure Monitor and an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals, and the average of the three measurements will be used.
Systolic and Diastolic blood pressure in mmHg | 60 days
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken using an Omron IntelliSense® Blood Pressure Monitor and an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals, and the average of the three measurements will be used.
Systolic and Diastolic blood pressure in mmHg | 90 days
  After the subject has rested for five minutes in a sitting position, blood pressure measurements will be taken using an Omron IntelliSense® Blood Pressure Monitor and an arm cuff suitable for the body size. Three readings will be taken at five-minute intervals, and the average of the three measurements will be used.
Body composition and body fat percentage | Baseline
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using an Inbody 770 (EUA)
Body composition and body fat percentage | 30 days
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using an Inbody 770 (EUA)
Body composition and body fat percentage | 60 days
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using an Inbody 770 (EUA)
Body composition and body fat percentage | 90 days
  Body composition (fat and lean body mass) will be measured by bioelectric impedance using an Inbody 770 (EUA)
Periodic dietary record forms (24h record) | Baseline
  Periodic records will be completed by participants and reviewed by the nutritionist to check for any missing information (number of meals, added sugar, spoon size, quantity consumed, and type of preparation).
Periodic dietary record forms (24h record) | 30 days
  Periodic records will be completed by participants and reviewed by the nutritionist to check for any missing information (number of meals, added sugar, spoon size, quantity consumed, and type of preparation).
Periodic dietary record forms (24h record) | 60 days
  Periodic records will be completed by participants and reviewed by the nutritionist to check for any missing information (number of meals, added sugar, spoon size, quantity consumed, and type of preparation).
Periodic dietary record forms (24h record) | 90 days
  Periodic records will be completed by participants and reviewed by the nutritionist to check for any missing information (number of meals, added sugar, spoon size, quantity consumed, and type of preparation).
Body Mass Index (BMI) | Baseline
  Weight in kg and height in meters will be used to calculate BMI
Body Mass Index (BMI) | 30 days
  Weight in kg and height in meters will be used to calculate BMI
Body Mass Index (BMI) | 60 days
  Weight in kg and height in meters will be used to calculate BMI
Body Mass Index (BMI) | 90 days
  Weight in kg and height in meters will be used to calculate BMI
Waist circumference in centimeters | Baseline
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (midway between the 10th rib and the iliac crest), as recommended by the World Health Organization, and hip circumference over the widest point over the buttocks to the nearest centimeter.
Waist circumference in centimeters | 30 days
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (midway between the 10th rib and the iliac crest), as recommended by the World Health Organization, and hip circumference over the widest point over the buttocks to the nearest centimeter.
Waist circumference in centimeters | 60 days
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (midway between the 10th rib and the iliac crest), as recommended by the World Health Organization, and hip circumference over the widest point over the buttocks to the nearest centimeter.
Waist circumference in centimeters | 90 days
  A certified non-stretch tape measure will be used to measure waist circumference (WC) at the natural waist (midway between the 10th rib and the iliac crest), as recommended by the World Health Organization, and hip circumference over the widest point over the buttocks to the nearest centimeter.
Height in centimeters | Baseline
  Height will be measured to the nearest 0.1 cm using a certified stadiometer
Height in centimeters | 30 days
  Height will be measured to the nearest 0.1 cm using a certified stadiometer
Height in centimeters | 60 days
  Height will be measured to the nearest 0.1 cm using a certified stadiometer
Height in centimeters | 90 days
  Height will be measured to the nearest 0.1 cm using a certified stadiometer
Blood sample | Baseline
  blood: collection after 12 hours of fasting, with evaluation of lipid profile (total cholesterol, triglycerides, low-density LDL cholesterol, high-density HDL cholesterol, very low-density VLDL cholesterol), blood glucose, glycated hemoglobin (HbA1c), inflammatory markers C-reactive protein (CRP-T) and tumor necrosis factor (TNF).
Blood sample | 90 days
  blood: collection after 12 hours of fasting, with evaluation of lipid profile (total cholesterol, triglycerides, low-density LDL cholesterol, high-density HDL cholesterol, very low-density VLDL cholesterol), blood glucose, glycated hemoglobin (HbA1c), inflammatory markers C-reactive protein (CRP-T) and tumor necrosis factor (TNF).
Genetic Analysis | 90 days
  Using the Real Time Polymerase Chain Reaction (real-time PCR) system on Step One PlusTM equipment

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrindo Ideais Research Center, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2025-04-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT06978504/ICF_000.pdf